CLINICAL TRIAL: NCT01710735
Title: Skeletal Muscle Contractility, Self-reported Pain and Tissue Sensitivity in Females With Neck/Shoulder Pain and Upper Trapezius Myofascial Trigger Points- a Randomized Intervention Study
Brief Title: Skeletal Muscle Contractility, Self-reported Pain and Tissue Sensitivity in Females With Neck/Shoulder Pain and Trapezius MFTrPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Lundbeck Foundation (Other); Dansk Kiropraktor Fond (Unknown); IMK Almene Fond (Other)
Responsible Party: Principal Investigator, Corrie Myburgh, Dr, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Muscle and needling
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Myofascial Pain Syndrome
Keywords: TP; Myofascial pain
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry needling (deep) (Experimental): Subjects receive dry needle insertion deeper than 1,5cm below the skin of the Trapezius.
  Interventions: Procedure: Dry needling
- Dry needling (superficial) (Active Comparator): Insertion of dry needle less than 1cm.
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Dry needling — Insertion of acupuncture needle into a myofascial trigger point.
  Other Names: Acupuncture

SUMMARY:
In relation to Myofascial Triggerpoints (MFTrPs) of the upper Trapezius, this study will explore muscle contractility characteristics, the occurrence of post-intervention muscle soreness and the effect of dry needling on muscle contractile characteristics and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A clinically relevant MFTrP of the upper Trapezius musculature
* Self-reported pain of ≥3 on an eleven-point numerical pain rating scale (NRS-101).
* BMI less than 31

Exclusion Criteria:

* a history of chronic, systemic pathology (e.g. hemophilia)
* pre-existing neck/shoulder pathology/surgical procedures,
* clinical depression
* health-related legal action
* pregnant
* anti-inflammatory and/or chronic pain medication
* had received dry needling for a shoulder/neck disorder within 6 months prior to the study (to raise the level of patient naiveté) suffered from needle phobia

Ages: 20 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
muscle contractility | 30 minutes
  Measurements of maximal isometric muscle force (Fmax), and rate of force development (RDF)

SECONDARY OUTCOMES:
pressure-pain threshold | 60 seconds
  Algometer measurement of pressure-pain perception
NRS-101 | 60 seconds
  Self-reported pain

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hartvigsen Hartvigsen, PhD, Study Director — Univ. of Southern Denmark; Per Aagaard, PhD, Study Director — Univ. of Southern Denmark
Locations (1):
- Univ. of Southern Denmark, Odense, Funen, Denmark

REFERENCES:
- [Derived] Myburgh C, Hartvigsen J, Aagaard P, Holsgaard-Larsen A. Skeletal muscle contractility, self-reported pain and tissue sensitivity in females with neck/shoulder pain and upper Trapezius myofascial trigger points- a randomized intervention study. Chiropr Man Therap. 2012 Nov 25;20(1):36. doi: 10.1186/2045-709X-20-36. PMID 23176709
- [Derived] Hofer KA, Ruonala R, Albert VA. The double-corolla phenotype in the Hawaiian lobelioid genus Clermontia involves ectopic expression of PISTILLATA B-function MADS box gene homologs. Evodevo. 2012 Nov 1;3(1):26. doi: 10.1186/2041-9139-3-26. PMID 23116179